CLINICAL TRIAL: NCT02575144
Title: GEM-CLARIDEX: Lenalidomide and Dexamethasone (Ld) Versus Clarithromycin / Lenalidomide [Revlimid®] / Dexamethasone (BiRd) as Initial Therapy in Multiple Myeloma
Brief Title: GEM-CLARIDEX: Ld vs BiRd
Acronym: GEM-CLARIDEX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PETHEMA Foundation (Other)
Collaborators: Cabyc, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM-CLARIDEX
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Clarithromycin; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BiRd (Experimental): Subjects on the BiRD arm will receive clarithromycin, Revlimid (lenalidomide), and dexamethasone in 28-day cycles. Dosing is as follows:
  * Clarithromycin 500mg PO twice daily on days 1-28 for a 28-day cycle.
  * Lenalidomide 25mg PO daily on days 1-21 of a 28-day cycle for patients with a calculated creatinine clearance of >60 cc/min. Patients with a calculated creatinine clearance of <60 cc/min will receive 15 mgs PO daily on days 1-21 of a 28 cycle.
  * Dexamethasone 40mg PO will be given on days 1, 8, 15, 22 of a 28-day cycle.
  Interventions: Drug: Clarithromycin; Drug: Lenalidomide; Drug: Dexamethasone
- Rd (Active Comparator): Subjects on the Rd arm will receive Revlimid, and dexamethasone in 28-day cycles. Dosing is as follows:
  * Lenalidomide 25mg PO daily on days 1-21 of a 28-day cycle. If a dose of lenalidomide is missed, it should be taken as soon as possible on the same day. If it is missed for the entire day, it should not be made up. Vomited doses will not be made up.Patients with renal failure will recived an ajusted dose.
  * Dexamethasone 40mg PO will be given on days 1, 8, 15, 22 of a 28-day cycle. Missed or vomited doses will not be made up. If subject cannot tolerate oral dexamethasone, it will be given intravenously. In patients over 75 years old, dexametasona oral will be given at dose of 20mg on days 1, 8, 15, 22 .
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Clarithromycin — 500mg PO twice daily on days 1-28 for a 28-day cycle
  Arms: BiRd
Drug: Lenalidomide — 25mg PO daily on days 1-21 of a 28-day cycle for patients with a calculated creatinine clearance of >60 cc/min
Drug: Dexamethasone — 40mg PO will be given on days 1, 8, 15, 22 of a 28-day cycle

SUMMARY:
This phase III study, open-label, randomized study investigating lenalidomide and dexamethasone with and without biaxin in subjects with newly diagnosed, previously untreated MM. Eligible subjects will be randomized in a 1:1 ratio to receive a regimen consisting of either biaxin, lenalidomide, and low-dose dexamethasone (BiRd arm), or lenalidomide and low-dose dexamethasone (Rd arm). 306 patients will be included (50% in Spain (153) and 50% in the USA (153)

DETAILED DESCRIPTION:
BiRd Arm

Subjects on the BiRD arm will receive clarithromycin, Revlimid (lenalidomide), and dexamethasone in 28-day cycles. Dosing is as follows:

* Clarithromycin 500mg PO twice daily on days 1-28 for a 28-day cycle. If a dose of clarithromycin is missed, it should be taken as soon as possible on the same day. If it is missed for the entire day, it should not be made up. Vomited doses will not be made up.
* Lenalidomide 25mg PO daily on days 1-21 of a 28-day cycle for patients with a calculated creatinine clearance of >60 cc/min. Patients with a calculated creatinine clearance of <60 cc/min will receive 15 mgs PO daily on days 1-21 of a 28 cycle. If a dose of lenalidomide is missed, it should be taken as soon as possible on the same day. If it is missed for the entire day, it should not be made up. Vomited doses will not be made up.
* Dexamethasone 40mg PO will be given on days 1, 8, 15, 22 of a 28-day cycle. Missed or vomited doses will not be made up. If subject cannot tolerate oral dexamethasone, it will be given intravenously.

Rd Arm

Subjects on the Rd arm will receive Revlimid, and dexamethasone in 28-day cycles. Dosing is as follows:

* Lenalidomide 25mg PO daily on days 1-21 of a 28-day cycle for patients with a calculated creatinine clearance of >60 cc/min. Patients with a calculated clearance of <60 cc/min will receive 15 mgs PO daily on days 1-21 of a28 cycle. If a dose of lenalidomide is missed, it should be taken as soon as possible on the same day. If it is missed for the entire day, it should not be made up. Vomited doses will not be made up.
* Dexamethasone 40mg PO will be given on days 1, 8, 15, 22 of a 28-day cycle. Missed or vomited doses will not be made up. If subject cannot tolerate oral dexamethasone, it will be given intravenously.

Correlative studies: Relative dose intensity: Projected total dose per cycle of each component of assigned drug will be divided by the actual dose received and a ratio will be assessed for each cycle delivered.

MRD: Minimal residual disease testing will be performed in subjects who achieve complete response. MRD testing may be performed either by flow cytometry or polymerase chain reaction (PCR), whichever is more readily available at the study institution.

Subjects will continue their randomized treatment assignment until disease progression or unacceptable toxicity (whichever occurs first). In case toxicity precludes dosing of one agent (i.e dexamethasone, clarithromycin, lenalidomide), treatment regimen will continue with the remaining agents. Subjects unable to receive ALL the components of the assigned treatment arms will be removed from study after reasonable attempts to dose reduce and manage side effects. Subjects can also be removed from study at investigator's discretion, or if they withdraw consent. At completion or early discontinuation of treatment, subjects will be followed for 30 additional days or up to the initiation of subsequent treatment (whichever occurs first), after which they will be off the active treatment phase of the study. Long-term follow-up for disease status and survival will proceed until the subject has withdrawn consent, is lost to follow-up, or has died.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily sign and understand written informed consent
* Subject is >=65 years at the time of signing the consent form
* Subject has histologically confirmed MM that has never before been treated
* Subject has no prior anti-myeloma treatment therapy within 14 days prior to initiation of study treatment except for corticosteroids with a maximum allowed dosage equivalent to three pulses of dexamethasone (40mg daily for 4 days equals one pulse). Patients may have received prior adjuvant antiresorptive therapy (i.e., pamidronate or zoledronic acid) as routine care, or radiation therapy as palliation for pain and/or spinal cord compression
* Subject has measurable disease as defined by > 0.5 g/dL serum monoclonal protein, >10 mg/dL involved serum free light chain (either kappa or lambda) provided that the serum free light chain ratio is abnormal, >0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s) of at least 1cm in greatest dimension as measured by either CT scanning or MRI
* Subject has a Karnofsky performance status ≥60% (>50% if due to bony involvement of myeloma (see Appendix IV)
* Subject is able to take prophylactic anticoagulation as detailed in section 9.1 (patients intolerant to aspirin may use warfarin or low molecular weight heparin)
* If subject is a female of childbearing potential (FCBP), ( A female of childbearing potential is a sexually mature woman who:

  1. has not undergone a hysterectomy or bilateral oophorectomy; or
  2. has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). She must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with FCBP even if they have had a successful vasectomy. See Appendix III: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods
* Subject has a life expectancy ≥ 3 months
* Subjects must meet the following laboratory parameters:

  * Absolute neutrophil count (ANC) ≥750 cells/mm3 (1.0 x 109/L)
  * Hemoglobin ≥ 7 g/dL
  * Platelet count ≥ 75,000/mm3 (30 x 109/L if extensive bone marrow infiltration)
  * Serum SGOT/AST <3.0 x upper limits of normal (ULN)ç
  * Serum SGPT/ALT <3.0 x upper limits of normal (ULN)
  * Serum total bilirubin <2.0 mg/dL (34 µmol/L)

Exclusion Criteria:

* Subject has immeasurable MM (no measurable monoclonal protein, free light chains in blood or urine, or measureable plasmacytoma on radiologic scanning)
* Subject has a prior history of other malignancies unless disease-free for ≥ 5 years, except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or localized prostate cancer with Gleason score < 7 with stable prostate specific antigen (PSA) levels
* Subject has had myocardial infarction within 6 months prior to enrollment, or NYHA (New York Hospital Association) Class III or IV heart failure (see Appendix VI), Ejection Fraction < 35%, uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Female subject who is pregnant or lactating
* Subject has known HIV infection
* Subject has known active hepatitis B or hepatitis C infection
* Subject has active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program
* Subject is unable to reliably take oral medications
* Subject has known hypersensitivity to dexamethasone, clarithromycin, lenalidomide, or thalidomide
* Subject has a history of thromboembolic event within the past 4 weeks prior to enrollment
* Subject has any clinically significant medical or psychiatric disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent
* Subject has previously been treated for MM
* Patients with symptomatic primary amiloidosis or symptomatic secondary amiloidosis (in patients with diagnosis of múltiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Throught the study. Approximately 4 years

CONTACTS AND LOCATIONS:
Locations (26):
- Spain (26):
  - CHUAC, A Coruña
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Clinic, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital General de Castelló, Castelló
  - Hospital de Cabueñes, Gijón
  - Hospital Universitario Virgen de las Nieves, Granada
  - H. del SAS de Jerez, Jerez de la Frontera
  - Hospital de León, León
  - H. U. Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Costa del Sol, Marbella
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Univeristario Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - H. Clínico de Valencia, Valencia
  - Hospital Universitario Dr Peset, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - H. U. Txagorritxu, Vitoria-Gasteiz

REFERENCES:
- [Derived] Jelinek T, Bezdekova R, Zihala D, Sevcikova T, Anilkumar Sithara A, Pospisilova L, Sevcikova S, Polackova P, Stork M, Knechtova Z, Venglar O, Kapustova V, Popkova T, Muronova L, Chyra Z, Hrdinka M, Simicek M, Garces JJ, Puig N, Cedena MT, Jurczyszyn A, Castillo JJ, Penka M, Radocha J, Mateos MV, San-Miguel JF, Paiva B, Pour L, Rihova L, Hajek R. More Than 2% of Circulating Tumor Plasma Cells Defines Plasma Cell Leukemia-Like Multiple Myeloma. J Clin Oncol. 2023 Mar 1;41(7):1383-1392. doi: 10.1200/JCO.22.01226. Epub 2022 Oct 31. PMID 36315921
- [Derived] Puig N, Hernandez MT, Rosinol L, Gonzalez E, de Arriba F, Oriol A, Gonzalez-Calle V, Escalante F, de la Rubia J, Gironella M, Rios R, Garcia-Sanchez R, Arguinano JM, Alegre A, Martin J, Gutierrez NC, Calasanz MJ, Martin ML, Couto MDC, Casanova M, Arnao M, Perez-Persona E, Garzon S, Gonzalez MS, Martin-Sanchez G, Ocio EM, Coleman M, Encinas C, Vale AM, Teruel AI, Cortes-Rodriguez M, Paiva B, Cedena MT, San-Miguel JF, Lahuerta JJ, Blade J, Niesvizky R, Mateos MV. Lenalidomide and dexamethasone with or without clarithromycin in patients with multiple myeloma ineligible for autologous transplant: a randomized trial. Blood Cancer J. 2021 May 21;11(5):101. doi: 10.1038/s41408-021-00490-8. PMID 34021118
- See also: Pethema Foundation web — http://www.fundacionpethema.es/